CLINICAL TRIAL: NCT02466802
Title: Phase I Study of Regorafenib and Sildenafil for Advanced Solid Tumors
Brief Title: Study of Regorafenib and Sildenafil for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13-09812; HM20004297 (Other: IRB); NCI-2015-01101 (Registry Identifier: NCI)
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumor
Keywords: Advanced
MeSH Terms: interventions — regorafenib; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- A: regorafenib and sildenafil citrate (Experimental): Patients receive regorafenib and sildenafil citrate by mouth every day (PO QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Regorafenib; Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Regorafenib — Combination of regorafenib and of sildenafil when given to patients with advanced solid tumors. Regorafenib Administration and Treatment Schedule. Regorafenib will be taken orally once daily for the first 21 days of each 28-day cycle. Regorafenib will not be taken on the last 7 days of each cycle. Patients will be instructed as follows: Take regorafenib once daily with a low fat meal that contains less than 30% fat. Take the regorafenib tablets at about the same time each day. Swallow the tablets whole.
  Other Names: Stivarga; 755037-03-7; BAY 73-4506
Drug: Sildenafil Citrate — Combination of regorafenib and of sildenafil when given to patients with advanced solid tumors.Sildenafil Administration and Treatment Schedule. Sildenafil will be taken orally once daily at the same time the regorafenib dose is taken for the first 21 days of each 28-day cycle. Sildenafil will not be taken on the last 7 days of each cycle.
  Other Names: Viagra; SILDENAFIL; Revatio; 171599-83-0

SUMMARY:
This is a phase 1 study of sildenafil in combination with regorafenib in patients with progressive advanced solid tumors. A modified 3+3 dose escalation design will be conducted for the dose escalation of the treatment combination: additional patients will be enrolled at the MTD until a total of 12 patients have been treated at the MTD.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, phase 1 trial to determine the RP2D of the combination of regorafenib and sildenafil. Both study medications will be taken orally on days 1-21 of each 28-day cycle.

Using a modified 3+3 dose escalation design, 3-6 patients with an advanced solid tumor will be enrolled at each dose level. Additional patients will be enrolled at the MTD until a total of 12 patients have been treated at the MTD.

Eligible patients will have received available standard treatments. Patients with solid tumors for which regorafenib would be considered a standard treatment are eligible as long as regorafenib has not been previously administered.

Blood samples will be collected for correlative studies including PK, PD, and CTCs. Tumor samples archived from a previous biopsy or surgery will also be collected for correlative studies.

ELIGIBILITY:
Inclusion Criteria:

• Advanced solid tumor that has progressed during or after treatment with approved therapies or for which there is no standard effective therapy available

* Note: patients with solid tumors for which regorafenib would be considered a standard treatment are eligible as long as regorafenib has not been previously administered

  * Measurable or evaluable disease by RECIST v1.1
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
  * Absolute neutrophil count (ANC) >= 1500/mm^3
  * Platelets >= 100,000/mm^3
  * Hemoglobin > 9 g/dL (untransfused)
  * Creatinine =< 1.5 x upper limit of normal (ULN) for the laboratory or calculated or actual creatinine clearance >= 60 mL/min
  * Proteinuria =< grade 1 (ie, =< 1+ [30 mg/dL] using a random urine sample or < 1.0 gm using a 24-hour sample)
* Note: if urine sample indicates >= grade 2 proteinuria (ie, 2+ [100 mg/dL]), a 24-hour urine sample must be collected and tested; urine protein in the 24-hour sample must be < 1.0 gm/24 hours • Total bilirubin =< 1.5 x ULN for the laboratory
* Exception: if a patient has documented Gilbert's syndrome and a total bilirubin is > 1.5 x ULN, the total bilirubin requirement may be waived provided the direct bilirubin is within normal limits (WNL) for the laboratory

  * Aspartate aminotransferase (AST) =< 2.5 x ULN for the laboratory
  * Alanine aminotransferase (ALT) =< 2.5 x ULN for the laboratory
  * Alkaline phosphatase =< 2.5 x ULN for the laboratory (=< 5 x ULN for patients with cancer involving the liver and/or bone)
  * Non-hematologic toxicities from previous cancer therapies resolved to =< grade 1
  * International normalized ratio (INR) is =< 1.5
  * Activated partial thromboplastin time (aPTT) =< 1.5 x ULN for the laboratory
  * Left ventricular ejection fraction (LVEF) assessed by echocardiogram within 3 months prior to initiation of study treatment indicates an LVEF of >= 50%
  * A woman of childbearing potential (WCBP), defined as a woman who is < 60 years of age and has not had a hysterectomy, must have a documented negative serum pregnancy test within 7 days prior to initiating study treatment
  * A WCBP and a male patient with a partner who is a WCBP must agree to use a medically accepted method for preventing pregnancy for the duration of study treatment and for 2 months following completion of study treatment
  * Ability to understand and willingness to sign the consent form written in English
* Note: the consent form must be signed prior to the conduct of any trial-specific procedure

Exclusion Criteria:

* Meningeal metastases or brain metastases that are symptomatic or untreated * Note: patients who are asymptomatic and have had post-treatment imaging that indicates stable brain disease are eligible; (patients with meningeal metastasis are not eligible even if stable following treatment); also, note that brain imaging is required within 8 weeks prior to initiation of study therapy
* Any investigational agent within 4 weeks prior to initiating study treatment
* Previous therapy with regorafenib
* If sorafenib was previously administered, intolerance to sorafenib
* Inability to swallow medication
* Known or suspected malabsorption condition or obstruction
* Contraindications to sildenafil including:

  * Known retinitis pigmentosa
  * History of priapism related to PDE5 inhibitors (eg, sildenafil, vardenafil, tadalafil)
  * Presence of nonmalignant hematologic disorders, such as sickle cell disease, that may increase the risk of priapism
* Contraindication to antiangiogenic agents, including:

  * Serious non-healing wound, non-healing ulcer, or bone fracture
  * Major surgical procedure or significant traumatic injury within 4 weeks prior to initiating study treatment
  * Pulmonary hemorrhage/bleeding event >= grade 2 within 12 weeks prior to initiating study treatment
  * Any other hemorrhage/bleeding event >= grade 3 within 12 weeks prior to initiating study treatment
* History of organ allograft including corneal transplant
* Any documented history of thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or pulmonary embolism within 6 months prior to initiating study treatment

  * Note: patients with a tumor-associated thrombus of locally-involved vessels should not be excluded from participating in the study
* Evidence of bleeding diathesis or coagulopathy
* Resting systolic blood pressure (BP) < 100 mmHg
* Hypertension defined as systolic BP >= 140 mmHg or diastolic BP >= 90 mmHg despite optimal medical management
* Active or clinically significant cardiac disease including any of the following:

  * Unstable angina (eg, anginal symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
  * Myocardial infarction within 6 months prior to initiating study treatment
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers
  * New York Heart Association (NYHA) class III or IV congestive heart failure
* Seizure disorder requiring medication
* Serious (ie, >= grade 3) uncontrolled infection
* Known human immunodeficiency virus (HIV) seropositivity

  * Note: HIV testing is not required
* Chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Pleural effusion or ascites that causes respiratory compromise (ie, >= grade 2 dyspnea)
* Untreated or metastatic pheochromocytoma
* Planned ongoing treatment with other drugs thought to potentially have adverse interactions with either of the medications included in the study treatment, for example:

  * Alpha 1-blockers
  * Vasodilators, such as nitrates
  * Other PDE5 inhibitors, eg, vardenafil, tadalafil
  * Therapeutic anticoagulation with vitamin K antagonists (eg, warfarin), heparins and heparinoids, or direct thrombin inhibitors (DTIs) ** Note: prophylactic low-dose anticoagulation to maintain vascular access devices or low-dose daily aspirin for cardiac health is permitted
  * Immunosuppressants such as tacrolimus, leflunomide or tofacitinib, roflumilast, pimecrolimus

    ** Note: administration of steroids as part of symptom management or for other supportive care purposes is permitted
  * STRONG cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and/or STRONG CYP3A4 inducers ** Note: if such medications have been used, patients must have discontinued these agents >= 2 weeks prior to initiating study treatment
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
To determine the recommended phase 2 dose (RP2D) of the combination of regorafenib and of sildenafil when given to patients with advanced solid tumors. | 28 days
  Patients' treatment dosing level, dose modification, DLTs, and evaluability for DLTs will be listed and summarized by basic descriptive statistics (such as frequency and proportion). The MTD/RP2D will be found based on the Definitions of Dose-Limiting Toxicity, Maximum Tolerated Dose, and Recommended Phase 2 Dose. RP2D for the combination of regorafenib and sildenafil that is less than or the same as the MTD.

SECONDARY OUTCOMES:
To evaluate the safety and toxicity of the regorafenib and sildenafil combination | Up to 30 days after completion of study treatment
  Adverse events reported according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0. Adverse events (AEs) characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) to determine safety and toxicity of the combination of regorafenib and sildenafil.
To explore the antitumor effects of the regorafenib and sildenafil combination | Up to 30 days after completion of study treatment
  Tumor response based on Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
To determine the pre-treatment expression of phosphodiesterase type 5 (PDE5) in tumor samples | 12- 24 months
  Pre-treatment PDE5 expression identified by immunohistochemistry using archived tumor tissue. Pre-treatment PDE5 expression identified by immunohistochemistry (IHC) using archived tumor tissue.
To evaluate the impact of sildenafil on the pharmacokinetics of regorafenib | 12-24 months
  Regorafenib plasma concentration measured at a total of 6 time points: at baseline (pre-treatment) and at 5 time points in cycle 1. Plasma concentration of regorafenib measured at 6 time points: at baseline (pre-treatment) and in cycle 1 on day 1 (post-treatment), on day 15 (pre- and post-treatment), and on day 21 (pre- and post-treatment)

OTHER OUTCOMES:
To explore the PD relationships between regorafenib and tumor response | 12-24 months
  Quantity of total and free regorafenib measured by in vitro RAF-1 kinase activity inhibition using plasma samples collected at baseline (pre-treatment) and in cycle 1 (post-treatment on day 1, pre- and post-treatment on day 15, and pre- and post-treatment on day 21)
To assess the feasibility of isolating, enumerating, and analyzing CTCs to characterize cGMP within tumor cells | Up to 30 days after completion of study treatment
  Characteristics of cGMP found in CTCs isolated and enumerated using the ApoStream DEPfff enrichment device with blood samples collected at baseline (pre-treatment), on days 1 and 15 in cycle 1, and at the time of each tumor response assessment
To assess the bioactivity of sildenafil in plasma | 12-24 months
  Quantity of total sildenafil measured by elevated VASP-1 phosphorylation ex vivo using plasma samples collected at baseline (pre-treatment) and in cycle 1 (post-treatment on day 1, pre- and post-treatment on day 15, and pre- and post-treatment on day 21)
To assess the cytokine/growth factor levels in plasma | Up to day 21 of course 1
  Quantity of cytokines/growth factors measured using a Bio-Rad MAGPIX multiplex reader ex vivo using plasma samples collected at baseline (pre-treatment) and in cycle 1 (post-treatment on day 1, pre- and post-treatment on day 15, and pre- and post-treatment on day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Poklepovic AS, Gordon SW, Kothadia S, McGuire WP, Thacker LR, Deng X, Tombes MB, Shrader E, Hudson D, Bandyopadhyay D, Ryan AA, Kmieciak M, Smith S, Dent P. A phase 1 study of regorafenib and sildenafil in adults with advanced solid tumors. Anticancer Drugs. 2024 Jun 1;35(5):450-458. doi: 10.1097/CAD.0000000000001584. Epub 2024 Mar 8. PMID 38452059
- [Derived] Booth L, Roberts JL, Rais R, Cutler RE Jr, Diala I, Lalani AS, Hancock JF, Poklepovic A, Dent P. Neratinib augments the lethality of [regorafenib + sildenafil]. J Cell Physiol. 2019 Apr;234(4):4874-4887. doi: 10.1002/jcp.27276. Epub 2018 Sep 10. PMID 30203445